CLINICAL TRIAL: NCT04489940
Title: A Phase II, Multicenter, Open Label Study of Bintrafusp Alfa (M7824) Monotherapy in Participants With HMGA2-expressing Triple Negative Breast Cancer
Brief Title: Bintrafusp Alfa in High Mobility Group AT-Hook 2 (HMGA2) Expressing Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely discontinued by the sponsor due to probability of success which was too low to justify the continuation of recruitment.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS200647_0020; 2019-004833-18 (EudraCT Number)
Record Dates: First submitted 2020-07-27; First posted 2020-07-28 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: M7824; Bintrafusp alfa; Programmed death-ligand 1; Transforming growth factor-β (TGF-β); Breast Cancer; MS200647
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bintrafusp alfa (Experimental)
  Interventions: Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Bintrafusp alfa — Participants received an intravenous infusion of 1200 milligrams (mg) bintrafusp alfa once every 2 weeks until confirmed disease progression, unacceptable toxicity, study withdrawal or death.
  Other Names: M7824

SUMMARY:
The main purpose of this study was to evaluate bintrafusp alfa monotherapy in participants with triple negative breast cancer (TNBC) who express high levels of HMGA2 as determined by a centralized reverse transcriptase-polymerase chain reaction (RT-PCR) test.

ELIGIBILITY:
Inclusion Criteria:

* Study participants have histologically or cytologically confirmed TNBC
* Absence of human epidermal growth factor receptor 2 (HER2), estrogen receptor, and progesterone receptor expression must be documented (criteria for defining TNBC are outlined in the protocol)
* Participants must have received at least one line of systemic therapy for metastatic disease and have progressed on the line of therapy immediately prior to study entry. There is no limit to the number of prior therapies
* Participants may prescreen for HMGA2 expression while on preceding treatment, however screening should only occur if in the opinion of the Investigator, the participant would likely be eligible for study within 6 months
* Participants must have measurable disease
* Availability of either archival tumor tissue or fresh core or excisional biopsy of a tumor lesion (primary or metastatic, excluding bone biopsies) is mandatory to determine HMGA2 expression level prior to enrollment
* HMGA2 high tumor expression is required and will be determined by a central lab
* Participants who have Eastern Cooperative Oncology Group (ECOG) PS of 0 to 1
* Participants have a life expectancy greater than or equal to (>=) 12 weeks as judged by the Investigator at study start
* Participants have adequate hematological, hepatic and renal and coagulation function as defined in the protocol
* Participants with known Human Immunodeficiency Virus (HIV) infections are in general eligible if the criteria as defined in the protocol are met (Food and Drug Administration [FDA] Guidance on Cancer Clinical Trial Eligibility, March 2019)
* Participants with hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infections are in general eligible if the criteria as defined in the protocol are met (FDA Guidance on Cancer Clinical Trial Eligibility, March 2019)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention are excluded. Participants with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 4 weeks, and are not using steroids for at least 7 days prior to the start of study intervention
* Participants must not have received prior cancer treatment with any other immunotherapy or checkpoint inhibitors, or any other immune-modulating monoclonal antibody
* Participants that received any organ transplantation, including stem-cell transplantation, but with the exception of transplants that do not require immunosuppression
* Participants with significant acute or chronic infections
* Participants with active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Participants with clinically significant cardiovascular/cerebrovascular disease including: cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure, or serious cardiac arrhythmia
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (45):
- United States (15):
  - Medical Oncology Hematology Consultants, PA, Helen F. Graham Cancer Center, Suite 3400, Newark, Delaware
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - New York Oncology Hematology, P.C. - Albany, Albany, New York
  - TheOhio State University, Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - UPMC Hillman Cancer Center - Hillman Cancer Center, Monroeville, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - The West Clinic, Germantown, Tennessee
  - Texas Oncology, P.A. - Austin - Austin Central Cancer Center, Austin, Texas
  - Texas Oncology, P.A. - Medical City Dallas - Pediatric Hematology/Oncology, Dallas, Texas
  - Texas Oncology, P.A. - Plano, Plano, Texas
  - Texas Oncology-San Antonio Stone Oak, San Antonio, Texas
  - Texas Oncology, P.A. - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates - Hampton, Norfolk, Virginia
- Belgium (3):
  - Universitair Ziekenhuis Brussel - Geriatrie, Brussels
  - UZ Leuven, Leuven
  - AZ Sint-Maarten - PARENT, Mechelen
- France (6):
  - Centre François Baclesse - Pathologies Gynecologiques, Caen
  - Centre Léon Bérard, Lyon
  - Hôpital Privé du Confluent SAS, Nantes
  - Groupe Hospitalier Diaconesses - Hôpital De La Croix Saint Simon - service d'oncologie medicale, Paris
  - CARIO - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin
  - Institut Curie - Centre René Huguenin - Service d'Oncologie Médicale, Saint-Cloud
- Italy (7):
  - IEO Istituto Europeo di Oncologia, Milan
  - Ospedale San Raffaele, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale - Dipartimento di Senologia, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS - Oncologia Medica 2, Padua
  - Azienda Ospedaliero Universitaria Pisana - U.O. Oncologia II, Pisa
  - Policlinico Universitario Agostino Gemelli - UOC Oncologia Medica, Roma
  - Istituto Clinico Humanitas, Rozzano
- Russia (9):
  - SBIH of Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary" - Chemotherapy, Arkhangelsk
  - SBIH " Clinical Oncological Dispensary # 1" - Location, Krasnodar
  - SBIH " Clinical Oncological Dispensary 1" - Location, Krasnodar
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin" - Moscow Cancer Research Centre, Moscow
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - LLC "ClinicaUZI4D", Pyatigorsk
  - FSBI "Clinical Research and Practical Center for specialized medical care (oncology)", Saint Petersburg
  - Tomsk Research Instutite of Oncology - Chemotherapy, Tomsk
  - SBIH Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa
- Spain (5):
  - Hospital Universitario Reina Sofia - Dept of Oncology, Córdoba
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - Hospital Ruber Internacional - Servicio de Oncologia, Madrid
  - Hospital Universitario Ramon y Cajal - Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio - Servicio de Oncologia, Seville

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0020
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 participants were screened, of which 11 participants received bintrafusp alfa monotherapy.
Period: Overall Study
Arm/Group | Bintrafusp Alfa
Started | 11
Completed | 1
Not Completed | 10
Not completed — Other | 2
Not completed — Withdrawal by Subject | 2
Not completed — Death | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all participants, who were administered at least one infusion of bintrafusp alfa.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by an Independent Review Committee (IRC)
Description: The ORR was defined as the percentage of participants with a confirmed objective response of Complete Response (CR) or Partial Response (PR) according to RECIST v1.1 as assessed by IRC. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions.
Time Frame: Time from first study intervention up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response (DOR) According to RECIST Version 1.1
Description: DOR was defined for participants with a confirmed objective response as the time from first documentation of a confirmed objective response (CR or PR) according to RECIST 1.1 to the date of first documentation of objective PD or death due to any cause, whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by IRC.
Time Frame: From first documented objective response to PD or death due to any cause, assessed up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

3. Secondary Outcome: Durable Response Rate (DRR) of at Least 6 Months Assessed by an Independent Review Committee (IRC)
Description: DRR was defined as the number of participants having a DOR of at least 6 months, out of the total number of participants.
Time Frame: Time from first study intervention up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST Version 1.1 Assessed by the IRC
Description: PFS was defined as the time from first study intervention until the first documentation of PD or death due to any cause in the absence of documented PD, whichever occurred first. PD: At least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. The tumor response was determined according to RECIST version 1.1 and assessed by the IRC.
Time Frame: Time from first study intervention up to until the first documentation of PD or death, assessed up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by the Investigator
Description: DOR was defined for participants with a confirmed objective response as the time from first documentation of a confirmed objective response (CR or PR) according to RECIST 1.1 to the date of first documentation of objective PD or death due to any cause, whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in sum of longest diameter (SLD) of all lesions. PD: At least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by investigator.
Time Frame: From first documented objective response to PD or death due to any cause, assessed up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

6. Secondary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by the Investigator
Description: The ORR was defined as the percentage of participants with a confirmed objective response of Complete Response (CR) or Partial Response (PR) according to RECIST v1.1 as assessed by investigator. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions.
Time Frame: Time from first study intervention up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

7. Secondary Outcome: Durable Response Rate (DRR) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Investigator
Description: as for outcome 3
Time Frame: Time from first study intervention up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Investigator
Description: PFS was defined as the time from first study intervention until the first documentation of PD or death due to any cause in the absence of documented PD, whichever occurred first. PD: At least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. The tumor response was determined according to RECIST version 1.1 and assessed by the investigator.
Time Frame: Time from first study intervention up to the first documentation of PD or death, assessed up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of analysis are censored at the date of the last follow-up. OS was summarized by Kaplan-Meier (KM) methods.
Time Frame: Time from the first dose of study drug until occurrence of death due to any cause, assessed up to 321 days
Population: As per changes in planned analysis, the outcome measure related to efficacy were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Related AEs, and Adverse Events of Special Interest (AESIs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether considered related to the medicinal product or protocol-specified procedure. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAE was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious TEAEs and non-serious TEAEs. The AESIs considered in this study are infusion-related reactions including immediate hypersensitivity, immune-related adverse events, skin adverse events, bleeding events and anemia.
Time Frame: Time from first study intervention up to 321 days
Population: The Safety Analysis Set (SAF) analysis set included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: Count of Participants
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 11
Count of Participants
  Participants with TEAEs | 10
  Participants with Treatment-Related TEAEs | 5
  Participants with AESIs | 4

11. Secondary Outcome: Immediate Observed Serum Concentration at End of Infusion (Ceoi) of Bintrafusp Alfa
Description: Ceoi was the serum concentration observed immediately at the end of infusion. This was taken directly from the observed bintrafusp alfa concentration-time data.
Time Frame: Pre-dose, End of Infusion from Day 1 to 321
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

12. Secondary Outcome: Serum Trough Concentration Levels (Ctrough) of Bintrafusp Alfa
Description: Ctrough was the serum concentration observed immediately before next dosing.
Time Frame: Pre-dose, End of Infusion from Day 1 to 321
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) of Bintrafusp Alfa
Description: The detection of antibodies to bintrafusp alfa was performed using a validated ADA assay method with tiered testing of screening, confirmatory and titration.
Time Frame: Pre-dose, End of Infusion from Day 1 to 321
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetics were not assessed.
Arm/Group | Bintrafusp Alfa
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Time from first study intervention up to 321 days.
Arm/Group | Bintrafusp Alfa
All-Cause Mortality (participants affected / at risk) | 6/11
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bintrafusp Alfa (N=11)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pain (General disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Epilepsy (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bintrafusp Alfa (N=11)
Anaemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Ear pruritus (Ear and labyrinth disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Diverticulitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatine phosphokinase increase (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood phosphorus increased (Investigations) | 1
Blood thyroid stimulating hormone dec (Investigations) | 1
Blood urea increased (Investigations) | 1
C-reactive protein increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 1
Thyroxine free increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Respiratory tract infection viral (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Based on sponsors decision for early termination of the study due to lack of probability to achieve interim data allowing expansion of this study.

Hence, analysis for efficacy, or biomarker were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT04489940/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT04489940/SAP_001.pdf